CLINICAL TRIAL: NCT03434756
Title: Propioceptive StabilizerTM Training in the Abdominal Wall Muscles in Healthy Subjects: A Pilot Study
Brief Title: Stabilizer in Abdominal Wall Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Carlos Romero Morales, PhD, Universidad Europea de Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CIPI/087/17
Record Dates: First submitted 2018-02-06; First posted 2018-02-15 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Healthy
Keywords: ultrasound imaging; propioception; training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Propioceptive Training (Experimental)
  Interventions: Other: Propioceptive training of the abdominal wall muscles

INTERVENTIONS:
Other: Propioceptive training of the abdominal wall muscles — At the beginning, patients will be in a supine position, the lower edge of the StabilizerTM will be placed between the posterior superior iliac spines, aligned with the sacral base. Abdominal manoeuvre will be developed by the patients until they reach 40 mmHg and hold steadily for 10 seconds. Prior the examination, each subject practiced the abdominal manoeuvre three times with an ultrasound image feedback.

SUMMARY:
The aim of the study will be tried to observe if the propioceptive Stabilizer training is effective in abdominal wall muscles in healthy subjects. All the participants will be examined in two times. Initially, baseline measurements with ultrasound imaging will be taken without muscle activity. After, they will do the abdominal manoeuvre and it will take the ultrasound images.

DETAILED DESCRIPTION:
Inclusion criteria will be health participants with age between 18 to 45 years. Exclusion criteria were a BMI higher than 31 kg/m2, hypocapnia, any musculoskeletal condition in lumbopelvic region, skin and lower limb pathology (i.e., fracture, surgery).

Initially, baseline measurements will make following Whittaker et al. guidelines to measure thickness of the abdominal wall muscles (external oblique, EO; internal oblique, IO; transversus abdominis, TrA and rectus anterior, RA). All evaluations will be carry out by a single operator (B.M.P), who was a specialized physical therapist with 3 years of USI experience. A diagnostic ultrasound tool (Toshiba Aplio 500 Platinum, Toshiba American Medical Systems; CA, USA) with a 7 to 14-MHz-range linear transducer (18L7 PLT-1204BT type; 40-mm footprint) will be used for B mode ultrasound imaging. Ultrasound images of the EO, IO and TrAb muscles will be taken with the patients in supine position, with a cross reference point placed between the iliac crest and the inferior border of subcostal line, and the midaxilary line on the right side ; RA muscle was aligned with the umbilicus; and interrecti distance (IRD) will be measured just under the umbilicus. The measure for the thickness during the rest condition will be perform by the mean of 3 repeated values for each measure at the end of expiration, maintaining the transducer at the same point. Muscle thickness will be considered as the distance between the inside caliper lines of each muscle border. IRD will be described as the distance between the inside caliper lines of each RA muscles.

Once baseline measurements will be taken, the same measurements will make while the patients perform the exercise. This exercise specifically targets the abdominal wall muscles (EO, IO, TrA and RA). At the beginning, patients will be in a supine position, the lower edge of the StabilizerTM will be placed between the posterior superior iliac spines, aligned with the sacral base. Abdominal draw in maneuver (ADIM) was developed by the patients until they reach 40 mmHg and hold steadily for 10 seconds. Prior the examination, each subject will be practiced the ADIM three times with an ultrasound image feedback.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* Body mass index higher than 31 kg/m2,
* Hypocapnia,
* Any musculoskeletal condition in lumbopelvic region,
* Skin and lower limb pathology (i.e., fracture, surgery)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2018-02-18 (Actual); Primary Completion 2018-02-22 (Actual); Study Completion 2018-02-25 (Actual)

PRIMARY OUTCOMES:
Thickness abdominal wall muscles | 1 day
  The measure for the thickness during the rest condition will be perform by the mean of 3 repeated values for each measure at the end of expiration, maintaining the transducer at the same point. IRD will be only evaluated in the midline. Muscle thickness will be considered as the distance between the inside caliper lines of each muscle border. Interrecti distance will be described as the distance between the inside caliper lines of each Rectus Anterioris muscles.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Teyhen DS, Gill NW, Whittaker JL, Henry SM, Hides JA, Hodges P. Rehabilitative ultrasound imaging of the abdominal muscles. J Orthop Sports Phys Ther. 2007 Aug;37(8):450-66. doi: 10.2519/jospt.2007.2558. PMID 17877281
- [Background] Miura T, Yamanaka M, Ukishiro K, Tohyama H, Saito H, Samukawa M, Kobayashi T, Ino T, Takeda N. Individuals with chronic low back pain do not modulate the level of transversus abdominis muscle contraction across different postures. Man Ther. 2014 Dec;19(6):534-40. doi: 10.1016/j.math.2014.05.010. Epub 2014 Jun 20. PMID 25009124